CLINICAL TRIAL: NCT07131358
Title: Comparison of Efficacy of Three Preventive Methods to Reduce the Incidence of Coronal Caries in Mexican Schoolchildren: a Randomized Clinical Trial.
Brief Title: Comparison of the Efficacy of Three Preventive Methods to Reduce the Incidence of Coronal Caries in Schoolchildren
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Aida Borges, Aida Borges-Yañez, PhD, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UNAMexico CIE/0606/03/2025
Record Dates: First submitted 2025-08-09; First posted 2025-08-20 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Caries Prevention
Keywords: coronal caries; prevention; pit and fissure sealant; fluoride varnish
MeSH Terms: conditions — Van der Woude syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group conventional pit and fissure sealant (glass ionomer) plus fluoride varnish (Experimental): Participants receive application of glass ionomer pit and fissure sealant plus semestral applications of fluoride varnish to the first permanent molars, and dental health education program.
  Interventions: Device: Glass ionomer pit and fissure sealant plus fluoride varnish
- Group pit and fissure sealant with Giomer® technology (Experimental): Participants receive application of pit and fissure sealant with Giomer® technology to the first permanent molars, and dental health education program.
  Interventions: Device: Pit and fissure sealant with Giomer® technology
- Group fluoride varnish (Active Comparator): Participants receive semestral applications of fluoride varnish to the first permanent molars, and dental health education program.
  Interventions: Device: Fluoride varnish

INTERVENTIONS:
Device: Glass ionomer pit and fissure sealant plus fluoride varnish — Application of glass ionomer pit and fissure sealant plus fluoride varnish
  Arms: Group conventional pit and fissure sealant (glass ionomer) plus fluoride varnish
Device: Pit and fissure sealant with Giomer® technology — Application of pit and fissure sealant with Giomer® technology
  Arms: Group pit and fissure sealant with Giomer® technology
Device: Fluoride varnish — Biannual application of fluoride varnish
  Arms: Group fluoride varnish

SUMMARY:
The objective of this clinical trial is to compare the efficacy of three preventive methods in reducing the incidence of coronal caries in the first permanent molars of Mexican schoolchildren.

The main question to be answered is:

Which of the preventive methods (application of fluoride varnish (control group), application of a conventional pit and fissure sealant (glass ionomer) plus fluoride varnish, or application of a pit and fissure sealant with Giomer® technology) will be more effective in preventing coronal caries in the first permanent molars of Mexican schoolchildren?

Hypothesis: The incidence of coronal caries with the application of a conventional pit and fissure sealant (glass ionomer) plus fluoride varnish will be lower compared to the application of a pit and fissure sealant with Giomer® technology and compared to the application of fluoride varnish (control group).

Three groups will be formed (68 participants each): one group will receive the application of sodium fluoride varnish (control group), a second group will receive the application of conventional pit and fissure sealant (glass ionomer) plus sodium fluoride varnish, and a third group will receive the application of pit and fissure sealant with Giomer® technology.

All groups will receive dental health education (importance of oral health, information about dental caries, oral hygiene practices, and information about coronal caries prevention). Preventive agents will be administered according to the manufacturer's instructions. Clinical evaluations will be carried out at baseline 6, 12, 18 and 24 months. The incidence of coronal caries between groups will be compared with the presence of surfaces with progression of caries in the first permanent molars.

The best preventive method can be proposed for use in caries prevention programmes in schoolchildren. The results will provide elements for the dental surgeon in decision-making to prevent caries lesions in schoolchildren.

DETAILED DESCRIPTION:
Dental caries is one of the most prevalent diseases in children worldwide. Untreated dental caries has economic and social repercussions, can affect academic performance, and negatively impact quality of life. Because of this situation, the search for an effective and efficient preventive agent for coronal caries is very important.

Currently, it is not possible to establish which type of pit and fissure sealant is best in terms of efficacy for caries prevention in first permanent molars. The application of preventive agents with Giomer® technology appears to be a promising alternative compared to existing alternatives. However, there is very little scientific evidence regarding the efficacy of pit and fissure sealants with Giomer® technology for caries prevention and their relative efficacy compared to other types of sealants. Furthermore, the evidence is limited and inconclusive regarding the efficacy of pit and fissure sealant plus fluoride varnish compared to pit and fissure sealant alone.

The use of pit and fissure sealants in school-aged children and the promotion of self-care practices should be included in prevention programs. The large proportion of children with treatment needs at the state and national levels emphasizes the need for oral health programs to reduce the incidence and prevalence of caries, as rehabilitation costs represent a significant burden for both families and health systems.

Hypothesis: The incidence of coronal caries in permanent first molars with the application of a conventional pit and fissure sealant (glass ionomer) plus fluoride varnish will be lower compared to the incidence of coronal caries in permanent first molars with the application of a pit and fissure sealant using Giomer® technology, and compared to the incidence of coronal caries in permanent first molars with the application of fluoride varnish (control group) after 24 months of follow-up.

General objective:

To compare the efficacy of three preventive methods in reducing the incidence of coronal caries in the first permanent molars of Mexican schoolchildren aged 6 to 8 years, in conjunction with an oral health education program, during a 24-month follow-up.

Specific objectives:

* To identify which of the three groups (fluoride varnish application (control group), application of a conventional sealant (glass ionomer) plus fluoride varnish application, or pit and fissure sealant with Giomer® technology) has the lowest incidence of dental caries in the permanent first molars of schoolchildren aged 6 to 8 years in the Municipality of Nezahualcóyotl, State of Mexico; during a 24-month follow-up.
* To identify if there is a difference between the retention rate of the conventional pit and fissure sealant (glass ionomer) with the retention rate of the self-etching pit and fissure sealant (Giomer®), during a 24-month follow-up.
* To identify if there are changes in the knowledge, attitudes, and practices of Mexican schoolchildren and their parents, before and after the application of the oral health education program.
* To identify if there are differences in the percentage of dental biofilm in Mexican schoolchildren after the application of the oral health education program.

METHODS Area: clinical research. Study type: Intervention. Study design: randomized controlled clinical trial. Study characteristics: prospective, longitudinal, comparative. Participant allocation: randomized. Study classification: efficacy study. Intervention model: parallel groups. Masking: blind (participant). Main purpose: Prevention. Study population: Schoolchildren aged 6 to 8 years attending public primary schools in the Municipality of Nezahualcóyotl, State of Mexico: "Emiliano Zapata" Primary School, "Venustiano Carranza" Primary School, and "Belisario Domínguez" Primary School.

Sample size: Three groups of 68 schoolchildren are required, in a no probabilistic convenience sampling.

Preventive agents will be administered according to the manufacturer's instructions.

Control group: Semi-annual application of fluoride varnish to the first permanent molars.

Conventional pit and fissure sealant (glass ionomer) plus fluoride varnish: Application of glass ionomer pit and fissure sealant and biannual fluoride varnish application on the first permanent molars.

Pit and fissure sealant with Giomer® technology: Application of pit and fissure sealant with Giomer® technology on the first permanent molars.

Before data collection, parents will be invited to participate and provided with an informed consent form. All schoolchildren between 6 and 8 years old will be invited to participate. The informed consent form will be provided to them, explaining any questions that may arise regarding their participation in the study. Children who choose to participate will place their fingerprint on the informed consent form.

An interview will be conducted to collect a series of sociodemographic variables. An interview will be conducted with the schoolchildren and a questionnaire will be administered to the parents of the schoolchildren to assess their knowledge, attitudes, and practices regarding oral health.

Prior to the application of preventive agents, caries risk assessment will be performed using the CAMBRA (Caries Management by Risk Assessment) system. Students will be classified in one of three categories: low risk, medium risk or high risk for caries; however, only students with moderate or high risk will be included in the study.

An initial oral clinical examination by a standardized dentist will be performed to evaluate the presence of the four permanent molars, the presence of dental caries and the presence of dental biofilm. The clinical examination will be conducted in public primary schools using a portable dental unit and artificial light.

Once the participants are selected, they will be randomly assigned to one of three groups.

The assessments will be repeated at 6, 12, 18, and 24 months. The examiner will be standardized for coronal caries assessment using the International Caries Detection and Assessment System (ICDAS) and for dental biofilm assessment. Two independent standardized examiners, who will not be involved in the initial clinical oral examination and the application of preventive agents, will conduct follow-up assessments of dental caries incidence.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren between 6 and 8 years of age, of both sexes, with at least one erupted permanent first molar, healthy or with incipient caries (ICDAS codes 1 and 2), attending public primary schools in the State of Mexico located in the municipality of Nezahualcóyotl.
* Schoolchildren with a moderate or high risk of tooth decay according to the caries risk assessment.

Exclusion Criteria:

* Schoolchildren with the presence of incisor-molar hypomineralization or dental fluorosis.
* Schoolchildren with the presence of sealants of fissures and fissures or with a history of their placement in any of the first permanent molars.
* School children who have a disability that prevents them from performing the oral clinical examination or interview.
* Schoolchildren with allergies or suspected allergies to milk protein and its derivatives, methacrylate monomer and/or acetone.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 204 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of coronal caries lesions | 24 months
  New lesions with caries progression

CONTACTS AND LOCATIONS:
Locations (3):
- Mexico (3):
  - Primary School "Belisario Dominguez", Nezahualcóyotl, State of Mexico
  - Primary School "Emiliano Zapata", Nezahualcóyotl, State of Mexico
  - Primary School "Venustiano Carranza", Nezahualcóyotl, State of Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ismail AI, Pitts NB, Tellez M; Authors of International Caries Classification and Management System (ICCMS); Banerjee A, Deery C, Douglas G, Eggertsson H, Ekstrand K, Ellwood R, Gomez J, Jablonski-Momeni A, Kolker J, Longbottom C, Manton D, Martignon S, McGrady M, Rechmann P, Ricketts D, Sohn W, Thompson V, Twetman S, Weyant R, Wolff M, Zandona A. The International Caries Classification and Management System (ICCMS) An Example of a Caries Management Pathway. BMC Oral Health. 2015;15 Suppl 1(Suppl 1):S9. doi: 10.1186/1472-6831-15-S1-S9. Epub 2015 Sep 15. No abstract available. PMID 26391116
- [Background] Rashed T, Alkhalefa N, Adam A, AlKheraif A. Pit and Fissure Sealant versus Fluoride Varnish for the Prevention of Dental Caries in School Children: A Systematic Review and Meta-Analysis. Int J Clin Pract. 2022 Sep 20;2022:8635254. doi: 10.1155/2022/8635254. eCollection 2022. PMID 36263239
- [Background] Kashbour W, Gupta P, Worthington HV, Boyers D. Pit and fissure sealants versus fluoride varnishes for preventing dental decay in the permanent teeth of children and adolescents. Cochrane Database Syst Rev. 2020 Nov 4;11(11):CD003067. doi: 10.1002/14651858.CD003067.pub5. PMID 33142363
- [Background] Ng TC, Chu CH, Yu OY. A concise review of dental sealants in caries management. Front Oral Health. 2023 Apr 17;4:1180405. doi: 10.3389/froh.2023.1180405. eCollection 2023. PMID 37138858
- [Background] Ramamurthy P, Rath A, Sidhu P, Fernandes B, Nettem S, Fee PA, Zaror C, Walsh T. Sealants for preventing dental caries in primary teeth. Cochrane Database Syst Rev. 2022 Feb 11;2(2):CD012981. doi: 10.1002/14651858.CD012981.pub2. PMID 35146744
- [Background] Ahovuo-Saloranta A, Forss H, Walsh T, Nordblad A, Makela M, Worthington HV. Pit and fissure sealants for preventing dental decay in permanent teeth. Cochrane Database Syst Rev. 2017 Jul 31;7(7):CD001830. doi: 10.1002/14651858.CD001830.pub5. PMID 28759120